CLINICAL TRIAL: NCT01586533
Title: A Phase II Double-blind, Randomized, Comparator-controlled Study of the Safety and Efficacy of Zoenasa™ Rectal Gel (Mesalamine Plus N-acetylcysteine) in Subjects With Left-sided Ulcerative Colitis
Brief Title: Study of the Safety and Efficacy of Zoenasa® Versus Mesalamine Enema in Subjects With Left-Sided Ulcerative Colitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Altheus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZA-201
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Ulcerative Colitis; Left-sided Ulcerative Colitis; Distal Ulcerative Colitis
Keywords: ulcerative colitis; UC; left-sided ulcerative colitis; distal ulcerative colitis; Zoenasa; mesalamine; mesalazine; 5-ASA; 5-aminosalicylic acid; N-acetylcysteine; acetylcysteine; NAC; enema; rectal gel
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoenasa-1:4 (Experimental)
  Interventions: Drug: Zoenasa-1:4
- Mesalamine Enema (Active Comparator)
  Interventions: Drug: Mesalamine Enema

INTERVENTIONS:
Drug: Zoenasa-1:4 — Zoenasa Rectal Gel (4.0g mesalamine [5-ASA], 1.0g N-acetylcysteine [NAC]; 60ml)
  Arms: Zoenasa-1:4
Drug: Mesalamine Enema — Mesalamine Rectal Suspension Enema (4.0g mesalamine [5-ASA], 60ml)
  Arms: Mesalamine Enema

SUMMARY:
This double-blind, randomized, comparator-controlled Phase II study is designed to establish the safety and efficacy of Zoenasa Rectal Gel compared to mesalamine enema in subjects with left-sided ulcerative colitis, as measured by the modified ulcerative colitis disease activity index (UCDAI), over 6 weeks of treatment. In this study, two cohorts of subjects will receive either Zoenasa-1:4 (1.0g NAC; 4.0g 5-ASA) investigational drug enema therapy or comparator mesalamine enema (4.0g 5-ASA). The study will enroll subjects randomized equally into the 2 cohorts. Each cohort will enroll approximately 60 subjects. The two arms of the trial will be enrolled concurrently in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects are eligible if they are ≥ 18 years of age and ≤ 64 years.
* They have a documented history of idiopathic ulcerative colitis based on endoscopic and/or histologic findings involving the left side of the colon, with mild to moderate active disease.
* Eligible subjects will have a documented history of ulcerative colitis, and a modified UCDAI score of 4-10, inclusive, with a Physician's rating of disease score of 2 points or less (mild or moderate active ulcerative colitis), rectal bleeding score of 1 or more (based on subject diary), and mucosal appearance score (based on endoscopy) of 1 point or more at baseline.
* Laboratory data:

  * White blood cell count between 4.0 - 12.0 K/mm3
  * Platelet count: 150 - 500 K/mm3
  * Hemoglobin > 10.0 g/dL
  * Total bilirubin < 1.5 mg/dL
  * Aspartate aminotransferase < 100 u/dL
  * Alanine aminotransferase < 100 u/dL
  * Alkaline phosphatase < 250 u/dL
  * Blood urine nitrogen < 40 mg/dL
  * Creatinine < 1.5 mg/dL
* Satisfies one of the following:
* Female subjects of childbearing potential must have a negative urine pregnancy test at screening; surgically sterile, post-menopausal, abstinent, or patient or partner agree to use a medically appropriate form of birth control from screening to until 1 month after the last dose of study medication.
* Male subjects must be surgically sterile, abstinent, or patient or partner compliant with a contraceptive regimen from screening to until 1 month after the last dose of study medication.
* They are able to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

* They have documented history of proximal or universal ulcerative colitis, proctitis or active proctitis confined to 15cm or less from the anal verge.
* They demonstrate signs and symptoms of fulminant colitis, bowel stricture, toxic megacolon, an anticipated need for blood transfusion for gastrointestinal bleeding, or demonstrate evidence of peritonitis.
* They receive a Physician's rating of disease severity as part of the modified UCDAI of 3 (severe disease) or an aggregate score of 11 or greater.
* They have shown prior documented history of evidence of high grade dysplasia on biopsy from endoscopic examinations.
* Their stool contains enteric pathogens or Clostridium difficile toxins.
* They have a history of recurrent Clostridium difficile infection.
* They have prior history of biologic therapy within the previous 4 years.
* They have received systemic steroids or immunosuppressants within the previous 4 weeks.
* Treatment in the last 14 days that included antibiotic, antifungal, antiparasitic medications, or rectally administered steroids (e.g. Cortenema®) or mesalamine enema (Rowasa®).
* Treatment in the last 7 days that included mesalamine (5-ASA) via oral administration (e.g. Asacol®, Lialda®, balsalazide, etc).
* They have a history of cancer (defined as malignancy within 5 years except for squamous cell or basal cell cancers of the skin), asthma, or bronchospasm.
* Positive pregnancy test or lactating subjects.
* There is evidence of chemical substance abuse.
* They have had repeated anti-inflammatory drug treatment (longer than 3 days at doses that exceed those available without a prescription) within the previous 7 days (with exception of aspirin at doses of 325mg/day or less for prophylaxis of cardiac disease), or initiated new non-steroidal anti-inflammatory (NSAID) treatment within the last 30 days.
* They have a known allergy to N-acetylcysteine or mesalamine, or have a history of serious AEs related to their use (including, but not limited to pancreatitis or hepatitis).
* They have a history of failure to retain enemas.
* Other clinically significant diseases that could interfere with the protocol compliance appear. These would include clinically important hematological, renal, hepatic, metabolic, psychiatric, central nervous system (CNS), pulmonary or cardiovascular disease.
* Use of any investigational medication within the previous 90 days.
* Any condition which the study physician judges to preclude safe participation in the study or to confound the evaluation of the study outcome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change in modified UCDAI at 6 weeks | 6 weeks
  Change from baseline in the modified Ulcerative Colitis Disease Activity Index (modified UCDAI) score at the end of the 6 week treatment period of Zoenasa™ Rectal Gel compared with mesalamine

SECONDARY OUTCOMES:
Change in modified UCDAI at 3 weeks | 3 weeks
  Change from baseline in the modified Ulcerative Colitis Disease Activity Index (modified UCDAI) score at the end of the 3 week treatment period of Zoenasa™ Rectal Gel compared with mesalamine
Clinical and endoscopic remission rates at 6 weeks | 6 weeks
  Proportion of patients in clinical and endoscopic remission at 6 weeks compared to baseline
Clinical and endoscopic remission rates at 3 weeks | 3 weeks
  Proportion of patients in clinical and endoscopic remission at 3 weeks compared to baseline
Clinical improvement rate after 6 weeks | 6 weeks
Clinical improvement rate after 3 weeks | 3 weeks
Endoscopic improvement rate at 6 weeks | 6 weeks
Endoscopic improvement rate at 3 weeks | 3 weeks
Change from baseline in endoscopic appearance after 6 weeks | 6 weeks
Change from baseline in endoscopic appearance after 3 weeks | 3 weeks
Time to resolution of rectal bleeding | Up to 6 weeks
Relapse rates at 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - Digestive Disease Associates, Gainesville, Florida
  - Digestive Medical Associates, Hialeah, Florida
  - The Center for Gastrointestinal Disorders, Hollywood, Florida
  - Miami Gastroenterology Consultants P.A., Miami, Florida
  - South Medical Research Group, Miami, Florida
  - Gastroenterology of Naples, Naples, Florida
  - Advanced Gastroenterology Associates, Palm Harbor, Florida
  - Shafran Gastroenterology, Winter Park, Florida
  - Tri-County Research, Athens, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - The Atlanta Center for Gastroenterology, Decatur, Georgia
  - St. Josephs Candler Health System, Savannah, Georgia
  - NCH Medical Group, Arlington Heights, Illinois
  - Gastrointestinal Clinic of Quad Cities, Davenport, Iowa
  - Professional Research Network of Kansas, Wichita, Kansas
  - Clinical Trials Management of Louisiana, Metairie, Louisiana
  - Dr. Jason Bozdin, M.D., Berkley, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Gregory Cammel, MD PLC, Wyoming, Michigan
  - GI Associates and Endoscopy Center, Jackson, Mississippi
  - Long Island Clinical Research Associates, Great Neck, New York
  - Research Associates of New York, New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - Carolina Digestive Health Associates, Davidson, North Carolina
  - LeBauer Research Associates, P.A., Greensboro, North Carolina
  - Greater Cincinnati Gastroenterology, Cincinnati, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Options Health Research, Tulsa, Oklahoma
  - Gastroenterology United Tulsa, Tulsa, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Houston Digestive Disease Clinic, Houston, Texas
  - Digestive Health Associates of Texas, Plano, Texas
  - Advanced Research Institute, South Ogden, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Digestive & Liver Disease Specialists, Norfolk, Virginia
  - Digestive Disease Institute, Seattle, Washington
  - Franciscan Research Center, Tacoma, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin